CLINICAL TRIAL: NCT00046488
Title: A Phase I Multicenter, Dose-Escalation Study of IDEC-152 (Anti-CD23 Monoclonal Antibody) in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Brief Title: Safety and Efficacy of IDEC-152 in the Treatment of Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Study MD, Biogen Idec
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 152-20
Record Dates: First submitted 2002-09-30; First posted 2002-10-02 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphoblastic Leukemia; Leukemia, Lymphoblastic, Chronic; Chronic Lymphocytic Leukemia; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — lumiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: IDEC-152 — 6 Dosing groups: 125mg/m2 weekly x 4, 250mg/m2 weekly x 4, 375mg/m2 weekly x 4, 500mg/m2 weekly x 4, 500mg/m2 3 times first week then weekly x 3, 500mg/m2 3 times per week x 4
  Other Names: Lumiliximab

SUMMARY:
To determine what side effects and what clinical effects if any the administration of this investigational product, IDEC-152 (an antibody against CD23 which is an important protein on leukemia cells and certain cells in the body's immune system), has on the CLL patient population.

ELIGIBILITY:
Inclusion Criteria:

* Signed IRB-approved informed consent.
* Greater than 18 years of age
* Proof of CD23+ CLL or small lymphocytic lymphoma (SLL)
* Progressive disease after at least 1 course of chemotherapy
* Acceptable hematologic status, liver function, renal function, and pulmonary function
* Patients of reproductive potential must agree to follow accepted birth control methods during treatment and for 3 months after completion of treatment

Exclusion Criteria:

* Previous exposure to IDEC-152 or other anti-CD23 antibodies
* Presence of HIV infection or AIDS
* Serious nonmalignant disease
* Active uncontrolled bacterial, viral or fungal infections.
* Clinically active autoimmune disease
* Pregnant or currently breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2002-09; Primary Completion 2004-04 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Determine a recommended Phase II dose for the treatment of patients with relapsed or refractory CLL | 48 months
Characterize the safety profile of IDEC-152 | 48 months

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics and pharmacodynamics of IDEC-152 in patients with relapsed or refractory CLL | 48 months
Evaluate the efficacy of IDEC-152 in patients with relapsed or refractory CLL | 48 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Research Site, La Jolla, California
  - Research Site, Baltimore, Maryland
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Columbus, Ohio
  - Research Site, Houston, Texas

REFERENCES:
- [Background] Byrd JC, O'Brien S, Flinn IW, Kipps TJ, Weiss M, Rai K, Lin TS, Woodworth J, Wynne D, Reid J, Molina A, Leigh B, Harris S. Phase 1 study of lumiliximab with detailed pharmacokinetic and pharmacodynamic measurements in patients with relapsed or refractory chronic lymphocytic leukemia. Clin Cancer Res. 2007 Aug 1;13(15 Pt 1):4448-55. doi: 10.1158/1078-0432.CCR-06-1463. PMID 17671129
- [Background] Pathan NI, Chu P, Hariharan K, Cheney C, Molina A, Byrd J. Mediation of apoptosis by and antitumor activity of lumiliximab in chronic lymphocytic leukemia cells and CD23+ lymphoma cell lines. Blood. 2008 Feb 1;111(3):1594-602. doi: 10.1182/blood-2007-03-082024. Epub 2007 Nov 21. PMID 18032710